CLINICAL TRIAL: NCT06925269
Title: Duchenne Muscular Dystrophy Quality of Life: Qualitative Interviews With Patients and Caregivers
Brief Title: DMD Voice: Qualitative Interviews With Patients and Caregivers
Status: Recruiting | Type: Observational
Sponsor: Red Nucleus Enterprise Solutions, LLC (Industry)
Collaborators: Italfarmaco S.A (Industry)
Responsible Party: Sponsor
Other Study IDs: CAS-ITF001-01
Record Dates: First submitted 2025-04-03; First posted 2025-04-13 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Duchenne Muscular Dystrophy (DMD)
Keywords: Duchenne; givinostat
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Subsample A - Caregivers: Caregivers of individuals with DMD treated with givinostat for at least 2 years
- Subsample A - Patients: Patients with DMD treated with givinostat for at least 2 years
- Subsample B - Caregivers: Caregivers of individuals with DMD never treated with givinostat

SUMMARY:
The purpose of this study is to understand DMD functional losses or abilities and their association with independence and quality of life from the perspective of individuals with DMD and/or and their caregivers.

This is a qualitative interview study in which individuals with DMD and/or their caregivers will be asked to participate in a semi-structured, approximately 60- minute interview. Interviews will focus on functional abilities and independence. Caregivers and boys with DMD will be interviewed. This study includes no treatment nor intervention; however, some participants are being treated by a drug that is approved in the U.S. and the U.K. and under investigation in other geographies.

ELIGIBILITY:
Inclusion Criteria:

Subsample A - Patients

Eligible participants for Subsample A must:

* Have been treated with Givinostat for at least 2 years
* Be at least 10 years of age with signed consent of a parent or legal guardian
* Be currently taking givinostat
* Willing and able to participate in a video and/or audio recorded interview

Subsample A - Caregivers

Eligible caregivers for Subsample A must:

* Be a parent or legal guardian of an individual with DMD that has been taking givinostat for at least two years
* Willing and able to participate in a video and/or audio recorded interview

Subsample B - Caregivers

Eligible caregivers for Subsample B must:

* Provide care to an individual with DMD who is unable to raise their hands above their head as confirmed by the caregiver
* Reside in the United States or Canada
* Able to read, speak, and understand English
* Willing and able to participate in a video and/or audio recorded interview Have access to a stable internet connection

Exclusion Criteria:

-

Min Age: 10 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Caregivers of individuals with Duchenne Muscular Dystrophy (DMD) and patients with DMD
Sampling Method: Non-Probability Sample
Enrollment: 68 (Estimated)
Dates: Start 2025-03-31 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Qualitative Interview | 60 minutes
  Participants will participate in a semi-structured interview

CONTACTS AND LOCATIONS:
Overall Officials: Mindy Leffler, M.Ed., Principal Investigator — Red Nucleus Solutions
Locations (1):
- Red Nucleus, Yardley, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No